CLINICAL TRIAL: NCT02770820
Title: Phase I/II Study of Autologous (Central Memory/Naïve) CD8+ T Cells That Have Been Transduced to Express a WT1-Specific T Cell Receptor for Treatment of AML
Brief Title: Laboratory-Treated (Central Memory/Naive) CD8+ T Cells in Treating Patients With Newly Diagnosed or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to funding difficulties
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9296; NCI-2016-00042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9296 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH); RG9216011 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-03-25; First posted 2016-05-12 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia; EBV-Positive Neoplastic Cells Present; HLA-A*0201 Positive Cells Present; Blasts Under 5 Percent of Bone Marrow Nucleated Cells; Elevated WT1
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (autologous CD8 T cells) (Experimental): Beginning 4 weeks after completion of last course of consolidation chemotherapy, patients receive autologous WT1-TCRc4 gene-transduced CD8+ TCM/TN lymphocytes IV over 1-4 hours on day 0 and again after a minimum of 3 weeks. Beginning 6 hours after the second infusion of T cells, patients also receive aldesleukin SC BID for 14 days in the absence of disease progression or unacceptable toxicity. Patients who have clinically benefitted from T cell therapy may receive additional infusions of T cells and aldesleukin at the discretion of the PI and the attending physician.
  Interventions: Biological: Aldesleukin; Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects of laboratory-treated (central memory/naive) cluster of differentiation 8+ T cells (autologous Wilms tumor [WT]1-T cell receptor [TCRc]4 gene-transduced CD8-positive central memory T-cells [TCM]/naive T cells [TN] lymphocytes) and how well it works in treating patients with acute myeloid leukemia that is newly diagnosed or has come back. Genetically modified therapies, such as autologous WT1-TCRc4 gene-transduced CD8-positive TCM/TN lymphocytes, are taken from a patient's blood, modified in the laboratory so they specifically may kill cancer cells with a protein called WT1, and safely given back to the patient. The "genetically modified" T-cells have genes added in the laboratory to allow them to recognize leukemia cells that express WT1 and kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety/potential toxicities associated with treating high-risk acute myeloid leukemia (AML) patients with autologous CD8+ T cells (polyclonal Tn and Tcm cells; Epstein-Barr virus-specific T cells [Tebv cells]) that have been genetically-modified to express a high affinity WT1-specific TCR (TCRC4).

II. Determine the feasibility of reproducibly treating high-risk AML patients with autologous CD8+ T cells (polyclonal TN and TCM cells; Tebv cells) that have been genetically-modified to express a high affinity WT1-specific TCR (TCRC4).

III. Determine and compare the in vivo persistence in blood and at the primary tumor site (e.g. bone marrow, chloroma) of transferred autologous CD8+ T cells (polyclonal TN and TCM cells; TEBV cells) that have been genetically-modified to express a high affinity WT1-specific TCR (TCRC4).

EXPLORATORY OBJECTIVES:

I. Determine whether adoptively transferred autologous TCRC4-transduced CD8+ cells have anti-tumor activity in patients with acute myeloid leukemia.

Ia. In patients with measurable minimal residual disease (MRD) at the time of infusion of TCRC4-transduced CD8+ cells, changes in leukemic tumor burden will be measured by morphology, flow cytometry, cytogenetics/fluorescence in situ hybridization (FISH) and/or molecular testing at baseline and after infusion of T cells.

Ib. In all patients (those with or without measurable tumor burden prior to T cell transfer, including patients who convert to MRD-negative status during consolidation), the probability of relapse, disease-free survival and overall survival of patients receiving TCRC4-transduced CD8+ cells will be compared with patients in the observation arm.

II. Determine and compare the migration to the primary tumor site of subsets of the adoptively transferred autologous TCRC4-transduced CD8+ T cells (polyclonal TN and TCM cells; TEBV cells).

III. Determine and compare the in vivo functional capacity of transferred polyclonal autologous TCRC4-transduced CD8+ TCM, TN cells and TEBV CD8+ cells.

OUTLINE:

Beginning 4 weeks after completion of last course of consolidation chemotherapy, patients receive autologous WT1-TCRc4 gene-transduced CD8+ TCM/TN lymphocytes intravenously (IV) over 1-4 hours on day 0 and again after a minimum of 3 weeks. Beginning 6 hours after the second infusion of T cells, patients also receive aldesleukin subcutaneously (SC) twice daily (BID) for 14 days in the absence of disease progression or unacceptable toxicity. Patients who have clinically benefitted from T cell therapy may receive additional infusions of T cells and aldesleukin at the discretion of the principal investigator (PI) and the attending physician.

After completion of study treatment, patients are followed up weekly for 4 weeks, at 2, 3, 6, and 12 months, and then annually for 14 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (non-M3) acute myeloid leukemia (AML)
* Patients must be >= 15 kg
* Patients or parents/legal guardian must be able to give informed consent
* Patients must be able to provide blood and marrow samples and to undergo the procedures required for this protocol
* Elevated expression of WT1 in pre-treatment bone marrow or peripheral blood by either of two methods:

  * Increased expression of WT1 determined if the number of copies of WT1 divided by the number of copies of ABL x 10^4 is > 250 for bone marrow, or > 50 for peripheral blood;
  * Demonstration of WT1 overexpression will be determined by immunohistochemical staining (IHC) in blasts as compared to adjacent normal myeloid and erythroid precursors, as determined by a Fred Hutchinson/Seattle Cancer Care Alliance pathologist
* Demonstration of disease response to induction chemotherapy, in that patients must have achieve a morphologic remission (marrow that is at least 10% cellular with < 5% blasts on morphologic review) after 1-2 induction cycles, regardless of minimal residual disease or incomplete hematologic recovery (CRi)/incomplete platelet recovery (CRp) status
* Determination of "high-risk" disease; subjects must meet one of the determinants of "high-risk disease", in terms of being at very high risk for relapse without allogeneic stem cell transplant, as per one of the follow criteria:

  * A designation of "adverse" risk disease at the time of diagnosis, as defined by cytogenetic and molecular abnormalities specifically outlined in the 2017 European LeukemiaNet (ELN) guidelines for diagnosis and management of AML; these patients will meet "high-risk" designation, regardless of minimal residual disease or CRi/CRp status
  * Relapsed leukemia; patients with cytogenetic or molecular classification other that adverse risk by ELN who go on to demonstrate disease relapse after a minimum duration of remission of 6 months, but who then attain a second complete remission with repeat induction chemotherapy; these patients will meet "high-risk" designation, regardless of minimal residual disease or CRi/CRp status
  * Minimal residual disease, as defined by having detectable disease by one of the following criteria, but otherwise being in morphologic remission

    * MRD by flow cytometry at any time after induction chemotherapy or during consolidation chemotherapy, when patients are otherwise classified as being in morphologic remission, and as defined by any abnormal myeloid blasts identified by flow cytometric analysis
    * Cytogenetic MRD, as defined by a disease-specific abnormal karyotype at any point in patients who are otherwise in morphologic remission
    * Molecular minimal residual disease (MRD) with one of the following markers, as specified below, in patients who are otherwise in morphologic remission:

      * A normalized copy number (NCN) of > 0.001 for CBFB/MYHI1 or a normalized copy number (NCN) of > 0.050 for AMLI/ETO (RUNXI/RUNX1T1) after at least 4 cycles of consolidation chemotherapy
      * A < 2 log reduction in either CBFB/MYH11 or AMLI/ETO (RUNX1/RUNX1T1) in the bone marrow at the time of post-induction disease restaging (immediately after 1-2 cycles of induction therapy)
    * CRi/CRp, as defined by neutrophil count < 1000/ul (CRi) and/or platelet count < 100,000/ul (CRp), but otherwise being in morphologic remission; in pediatric patients, a platelet threshold of < 80,000/ ul will be used, as per consensus pediatric response criteria
* Human leukocyte antigen (HLA)-A*02:01 expression must be present for patient to be on treatment arm, HLA-A*02:01 expression absent in patients designated to observation arm

ELIGIBILITY FOR APHERESIS/BLOOD COLLECTION:

• HLA-A*02:01 expression

ELIGIBILITY FOR TREATMENT WITH TCRC4-TRANSDUCED CD8+ CELLS

* Response to therapy and completion of at least one cycle of consolidation therapy, and with disease status meeting one of the aforementioned "high-risk" criteria at the time of post-induction disease restaging as already outlined above
* Hematologic recovery from induction and other post-remission therapy (absolute neutrophil count [ANC] > 200/ul, platelet count > 20,000/ul) at the time of the study intervention
* No plan for allogeneic stem cell transplantation within 3 months
* Elevated expression above baseline of WT1 in bone marrow or peripheral blood
* Additionally, patients treated in stage 1, cohort #3 must be Epstein-Barr virus (EBV) seropositive, given the inclusion of T cells derived from an EBV-specific subset in this group
* Continued morphologic remission (< 5% blasts in the marrow, no circulating blasts or known extramedullary relapse) within 6 weeks of receiving the study intervention (specified as T cell infusion for cohort 1, or the start of lymphodepleting chemotherapy for cohorts 2 and 3)
* ELIGIBILITY FOR OBSERVATION ARM
* The patient meets all of the eligibility criteria for enrollment, but lacks expression of HLA-A*0201 as is needed to be enrolled on the treatment arm and for apheresis

Exclusion Criteria:

* Active autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease, inflammatory bowel disease) in which possible progression during treatment would be considered unacceptable by the investigators
* Previous allogeneic hematopoietic cell transplant (HCT)
* Any condition or organ toxicity deemed by the principal investigator (PI) or the attending physician to place the patient at unacceptable risk for treatment on the protocol
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling or unable to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to enrollment and initiation of treatment
* Clinically significant and ongoing immune suppression including, but not limited to: systemic immunosuppressive agents such as cyclosporine or corticosteroids (at an equivalent dose of 0.5 mg prednisone/kg per day, or higher), chronic lymphocytic leukemia (CLL), uncontrolled human immunodeficiency virus (HIV) infection (untreated or detectable viral load within 3 months of enrollment)
* Acute promyelocytic leukemia (M3 leukemia, per French-American-British classification)

EXCLUSION FOR TREATMENT WITH TCRC4-TRANSDUCED CD8+ CELLS

* Unable to generate antigen-specific WT1-specific CD8+ T cells for infusions; however, if a lower than planned number of cells is available, the patient will have the option to receive the generated WT1-specific T cells
* Systemic steroids should be stopped 2 weeks before the start of treatment; topical and inhaled steroids are allowed
* Symptomatic and refractory central nervous system (CNS) leukemia
* Absolute neutrophil count (ANC) < 200/ul prior to treatment
* Platelets < 20,000/ul prior to treatment
* If a patient meets other treatment eligibility but otherwise demonstrates delayed or poor recovery of peripheral blood counts to the above neutrophil and/or platelet thresholds, then treatment with the T cell intervention will be allowed if:

  * Neutrophil and/or platelet counts remain below the thresholds after a period of at least 6 weeks from last systemic chemotherapy; OR neutrophil and/or platelet counts remain below the thresholds in the setting of a maintenance therapy, such as midostaurin; and
  * The patient has detectable leukemia (e.g. flow cytometry positive or MRD by FISH or molecular testing); and
  * The P.l. or treating physician documents that the likely cause of cytopenias is underlying disease as opposed to another cause (e.g. medication)
* Ongoing >= grade 3 cardiac, pulmonary, renal, gastrointestinal or hepatic toxicities according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 toxicity criteria
* Karnofsky performance status score (age >= 16 years) or Lansky play score (age < 16 years) =< 40%
* Medical or psychological conditions that, according to the PI, would make the patient unsuitable candidate for cell therapy
* Pregnancy or breast-feeding; women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test result within 14 days before the first dose of WT1-specific T cell infusions; woman of non-childbearing potential will be defined as being postmenopausal greater than one year or who have had a bilateral tubal ligation or hysterectomy; all recipients of WT1-specific T cells will be counseled to use effective birth control during participation in this study and for 12 months after the last T cell infusion
* Treatment with alemtuzumab or other T cell-depleting antibodies within 6 months of T cell therapy
* Documented new infection within 24 hours of T cell infusion, or concern for new infection as suggested by an oral temperature > 38.2 degrees Celsius (C) within 24 hours of T cell infusion

  * ln patients who have T cells delayed because of development of fever (oral temperature > 38.2 degrees C) and who subsequently become afebrile (38.2 degrees C or less) for 24 hours without a documented infection, T cells may be administered
  * ln patients with a documented new infection within 24 hours of planned T cell infusion, they may go on to receive T cells after administration of directed antibiotic therapy and if they subsequently remain afebrile (38.2 degrees C or less) for at least 24 hours, and if it is deemed clinically appropriate by the Pl
  * Pre-existing infections requiring chronic maintenance therapy (e.g. chronic hepatitis B virus [HBV] or treated bacterial infections) are not an exclusion for T cell infusion as long as patients are on appropriate antimicrobial therapy for at least 1 month (e.g. for chronic hepatitis B or C viral infection) and who remain afebrile and without symptomatic evidence for uncontrolled chronic infection within 24 hours of T cell infusion; patients should also have a negative HIV test by viral load within 3 months of treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chapuis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Autologous CD8 T Cells)
Started | 7
Completed | 4
Not Completed | 3
Not completed — Death | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Autologous CD8 T Cells)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 63.21 [51.07 to 74.15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Serious Adverse Event (SAE)
Description: Evidence and nature of toxicities will be measured according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.This is the number of participants who experienced at least one adverse event (SAE).
Time Frame: 12 months after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous CD8 T Cells)
Number analyzed (Participants) | 7
Participants | 0

2. Primary Outcome: Feasibility of Subsets
Description: Feasibility of generating TCR-transduced TN and TCM subsets for adoptive immunotherapy in a high-risk AML population. This is the proportion of subjects who sign the treatment consent, have a T cell product generated, and ultimately receive the study intervention.
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous CD8 T Cells)
Number analyzed (Participants) | 7
Participants | 6

3. Primary Outcome: Number of Participants Whose Treatment Resulted in TCRC4-transduced CD8+ Polyclonal TCM and TN Cell Persistence.
Description: Comparison of the relative frequencies and duration of persistence of adoptively transferred TCRC4-transduced CD8+ polyclonal TCM and TN cells, and of TCRC4-transduced TEBV CD8+ cells in blood and at the primary tumor site(s). This is the number of participants whose blood samples displayed TCRC4-transduced CD8+ polyclonal TCM and TN cell Persistence in follow up.
Time Frame: 12 months after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous CD8 T Cells)
Number analyzed (Participants) | 7
Participants | 0

4. Other Pre Specified Outcome: Relative Maintenance
Description: of functional capacity and potential acquisition of phenotypic characteristics associated with T cell exhaustion in transferred WT1+ cell populations TN compared to TCM compared to TEBV C4-transduced CD8+ cells: decrease in blast counts in blood or marrow (by morphology and flow cytometry), and/or decrease in disease burden as detected by cytogenetics/FISH or molecular testing
Time Frame: Up to 15 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patients With or Without Detectable MRD
Description: comparison of probability of relapse, disease-free survival (DFS) and overall survival (OS) to patients in the observation arm
Time Frame: Up to 15 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Relative Frequencies at Primary Tumor Sites
Description: of TCRC4-transduced CD8+ polyclonal TCM and TN cells and EBV-specific (TEBV) cells compared to peripheral blood
Time Frame: Up to 15 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Relative Maintenance of Functional Capacity
Description: and potential acquisition of phenotypic characteristics associated with T cell exhaustion in transferred WT1+ cell populations TN compared to TCM compared to TEBV
Time Frame: Up to 15 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Treatment (Autologous CD8 T Cells)
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Autologous CD8 T Cells) (N=7)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (10)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02770820/Prot_SAP_000.pdf